CLINICAL TRIAL: NCT00759863
Title: LifeZig System for Individuals With Alzheimer's Disease
Brief Title: LifeZig Personalized Reminiscence Video With Slideshows and Music for Individuals With Alzheimer's and Dementia
Acronym: Lifezig
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Photozig, Inc. (Industry)
Responsible Party: Bruno Kajiyama, Photozig, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pz-A102b; R44AG022261 (NIH)
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Results first posted 2010-02-23 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-02

CONDITIONS: Alzheimer's Disease; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia

ARMS (2):
- Lifezig (Experimental): Subjects watch personalized reminiscence video channels developed by program staff with the help of family members/caregivers (using the LifeZig system)
  Interventions: Behavioral: Lifezig
- Usual Care (No Intervention): Subjects follow routine activities applied by nurses or caregivers, such as traditional reminiscence, crafts, singing, recreational activities, and other activities.

INTERVENTIONS:
Behavioral: Lifezig — Personalized Reminiscence Video
  Other Names: LifeZig Personalized Reminiscence Slideshow
  Arms: Lifezig

SUMMARY:
The LifeZig Project is a research study of a new reminiscence activity for individuals with Alzheimer's Disease (AD) and other types of dementia, based on the LifeZig system, with personalized video channels containing old photographs and music on television.

The goal of the LifeZig study is to enhance the quality of life for dementia patients and their families/caregivers, decrease the burden of care, and contribute to positive interaction between dementia patients and families/caregivers.

DETAILED DESCRIPTION:
This program creates personalized TV channels with old photographs of AD patients, music, narration and relaxing sounds; as an activity to relax dementia patients.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for dementia patients:

  * documented diagnosis of probable Alzheimer's or other type of dementia, medically stable, and visual/hearing capabilities to watch television.
* Inclusion criteria for family members/caregivers:

  * provide care or be a family member of dementia patient, have knowledge of the person, and be able to provide old photographs of dementia patient.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2006-08; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Kajiyama, MS, Principal Investigator — Photozig, Inc.
Locations (1):
- Photozig, Inc., Moffett Field, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lifezig | Usual Care
Started | 144 | 98
Completed | 124 | 80
Not Completed | 20 | 18
Not completed — Death, moved, or lost contact | 20 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lifezig | Usual Care | Total
Number analyzed (Participants) | 144 | 98 | 242
Age Continuous [Mean (Standard Deviation); unit: years] | 84.02 (7.31) | 84.48 (7.03) | 84.21 (7.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 80 | 196
  Male | 28 | 18 | 46
Region of Enrollment [Number; unit: participants]
  United States | 144 | 98 | 242

OUTCOME MEASURES:

1. Primary Outcome: Multidimensional Observation Scale for Elderly Subject
Description: This scale reflects the overall well-being of dementia patients. The construct being assessed is the quality of life of dementia patients, related to patient functioning, disoriented behavior, depression/anxiety, irritable behavior, and withdrawn behavior, consisting of 32 items, divided in four sub-scales: "Personal Care", "Communication, Awareness & Memory", "Mood", and "Interpersonal Awareness Behaviors". The overall score provides an indication of the overall perceived well-being of the dementia patient. Best value = 32. Worst Value = 144.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lifezig | Usual Care
Number analyzed (Participants) | 124 | 80
Units on a scale | 69.75 (19.05) | 77.99 (15.17)

2. Secondary Outcome: Revised Memory and Behavior Problems Checklist
Description: This scale measures the type/number of dementia patients disturbing behaviors, and how much they bother caregivers with 24 items describing possible troublesome behaviors that the patient might evidence in the past month. Caregivers are first asked whether the dementia patient had displayed any of these in the time period, and secondly to rate on a 5-point scale (0=not at all; 4= extremely) how much this "bothered or upset" them. A "conditional bother" score is calculated which is the "upset" or "bother" ratings for only the problematic behavior that occurred. Best value = 0. Worst Value = 96.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lifezig | Usual Care
Number analyzed (Participants) | 124 | 80
Units on a scale | 11.39 (10.82) | 15.55 (11.66)

3. Secondary Outcome: Center for Epidemiologic Studies Depression Scale
Description: The Center for Epidemiological Studies Depression scale (CES-D) is a 20-item measure that asks about the frequency of depressive symptoms (affective, psychological, and somatic) within the past week. The construct being assessed is the caregiver depression. Best value = 0. Worst Value = 60.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lifezig | Usual Care
Number analyzed (Participants) | 124 | 80
Units on a scale | 11.00 (8.35) | 10.43 (8.74)

ADVERSE EVENTS:
Arm/Group | Lifezig | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/144 | 0/98
Other Adverse Events (participants affected / at risk) | 0/144 | 0/98

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes